CLINICAL TRIAL: NCT07179835
Title: To Evaluate Periapical Healing Post Full Pulpotomy in Permanent Mandibular Teeth With and Without Apical Periodontitis
Brief Title: To Evaluate Periapical Healing Post Full Pulpotomy in Teeth With and Without Apical Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jigyasa Duhan
Record Dates: First submitted 2025-07-21; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- To evaluate success of full pulpotomy in mandibular permanent with apical periodontitis (Experimental): To evaluate success of full pulpotomy based on clinical and radiographic criteria in mandibular permanent with apical periodontitis
  Interventions: Procedure: Full pulpotomy in adults ≥18 years with restorable mandibular first or second molars diagnosed with irreversible pulpitis, with or without apical periodontitis.
- To evaluate success of full pulpotomy in mandibular permanent without apical periodontitis (Experimental): To evaluate and compare success of full pulpotomy based on clinical and radiographic criteria in mandibular permanent withoutapical periodontitis
  Interventions: Procedure: Full pulpotomy in adults ≥18 years with restorable mandibular first or second molars diagnosed with irreversible pulpitis, with or without apical periodontitis.

INTERVENTIONS:
Procedure: Full pulpotomy in adults ≥18 years with restorable mandibular first or second molars diagnosed with irreversible pulpitis, with or without apical periodontitis. — Comparison of full pulpotomy with MTA in teeth with and without apical periodontitis

SUMMARY:
This clinical study aims to evaluate the periapical and clinical healing outcomes of full pulpotomy using MTA in mandibular permanent molars diagnosed with symptomatic irreversible pulpitis. Patients will be stratified based on the presence or absence of apical periodontitis. Clinical and radiographic assessments will be conducted at baseline, 6 months, and 12 months to compare healing outcomes between groups. The study seeks to determine the effectiveness of full pulpotomy as a less invasive alternative to root canal treatment, even in teeth with apical pathosis.

DETAILED DESCRIPTION:
This prospective clinical study aims to evaluate the periapical and clinical healing outcomes of full pulpotomy using mineral trioxide aggregate (MTA) in mandibular permanent molars diagnosed with symptomatic irreversible pulpitis. Patients will be stratified based on the presence or absence of apical periodontitis. Clinical and radiographic assessments will be conducted at baseline, 6 months, and 12 months to compare healing outcomes between groups. The study seeks to determine the effectiveness of full pulpotomy as a less invasive alternative to root canal treatment, even in teeth with apical pathosis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient should be ≥18 years of age.
2. Restorable mature permanent 1st and 2nd Mandibular molars with extremely deep caries (≥2/3 dentine involvement)
3. Tooth should give positive response to pulp sensibility testing.
4. Radiographic finding of periapical index (PAI) score >/=3 (for test group) , score </= 2 (for control group)

Exclusion criteria

1. Teeth with immature roots.
2. No pulp exposure after caries excavation.
3. Bleeding could not be controlled in 10 minutes.
4. Signs of pulpal necrosis, sinus tract, swelling, insufficient bleeding after pulp exposure.
5. History of analgesic intake in previous 1 week, or antibiotic intake in 1 month.
6. Internal/external resorption.
7. Contributory medical history (alcoholism, smokers, diabetic, hypertension, drug dependency, Heart or valve disease, hepatitis, herpes, immunodeficiency (HIV), infectious diseases, kidney or liver, migraine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Success following complete pulpotomy | 12 MONTHS
  Clinical-Radiographic Success After Full Pulpotomy in Mandibular Molars With and Without Apical Periodontitis"

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No